CLINICAL TRIAL: NCT03955809
Title: Effects of İntraarticular and Periarticular Applied Drugs on Postoperative Pain Management in Artroscopic Knee Surgery for
Brief Title: Comparison the Effects of 3 Different Intraarticular Ketamine Doses on Postoperative Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, Associated Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: osagir3
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Arthroscopy
Keywords: Injection; Intra-Articular; arthroscopy; ketamine
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine 0.5 mg/kg (Active Comparator): ketamin 0.5 mg/kg intraarticular
  Interventions: Drug: Ketamine 0.5
- Ketamine 1 mg/kg (Active Comparator): ketamin 1 mg/kg intraarticular injection
  Interventions: Drug: Ketamine 1
- % 0.9 Saline (Sham Comparator): % 0.9 NaCL intraarticular injection
  Interventions: Drug: % 0.9 NaCl

INTERVENTIONS:
Drug: Ketamine 0.5 — İntrarticular Ketamine 0.5 mg/kg + 0.9 Nacl Total Volume 20 ml
  Other Names: Group 1
  Arms: Ketamine 0.5 mg/kg
Drug: Ketamine 1 — İntrarticular Ketamine 1 mg/kg + 0.9 NaCl Total Volume 20 ml
  Other Names: Group 2
  Arms: Ketamine 1 mg/kg
Drug: % 0.9 NaCl — Intraarticular %0.9 NaCl
  Other Names: Group 3
  Arms: % 0.9 Saline

SUMMARY:
the aim is to compare the effects of two different doses of intraarticular ketamine on postoperative pain scores and analgesic requirements.in knee artroscopy

DETAILED DESCRIPTION:
All pateints are going to be operated under general anesthesia. At the end of the study patients are going to be randomyl seperated into 3 groups. The surgeon is going the following drugs intraarticulary.

Group KL1: 0.5 mg/kg ketamin in % 0..9 NaCl at a total volume of 20 ml Group KL2: 1 mg/kg ketamin in % 0.9 NaCl at a total volume of 20 ml Group SL: 20 ml % 0.9 NaCl ll patients are going to receive a periarticula injection of 10 ml 0.5 bupivacaine and patient controlled analgesia with morphine.

VAS scores and total analgesic requirement is going to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Artroscopic surgery
* ASA I-II

Exclusion Criteria:

* Long time NSAID use
* Travmatic knee injury
* Long ter analgesic use
* Intraartiular catheter insertion at the end of surgery

Ages: 18 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain scores throughout time evaluated by VAS | VAS scores at rest and during activity will be evaluated for 24 hours. The first measurement will be recorded immediately after surgery and at 30 minutes interval for the first hour. Afterwards at 2.4.6.12.24.hours postoperatively.
  Pain scores are going to be evaluated by VAS scores at rest and VAS scores at activity
Difference in opioid Sparing effect measured through morphine amount delivered by a patient controlled analgesia device. | Total amount off delivered morphine will be recorded for 24 hours.
  The total amount of morphine delivered by the patient controlled analgesia device in the first 24 hours will be recorded.

SECONDARY OUTCOMES:
Time for discharge measured by eligible for discharge criteria | Discharge criterias will be evaluated every three hours until postoperative 24. hour. In patients who did not complete the discharge criteria in the postoperative 24 hours period, they will be defined as prolonged discharge.
  The time needed to fullfill the dicharge criteria (stable vital signs, able to walk, able to eat, nausea and vomit free, able to mixture)

IPD SHARING:
Plan to Share IPD: No